CLINICAL TRIAL: NCT06815029
Title: A Phase 1 Trial to Evaluate the Safety of IL13Rα2-Targeting Chimeric Antigen Receptor (CAR) T Cells With CRISPR Knockout of TGFβR2 in Patients With Recurrent or Progressive High-Grade Glioma (HGG)
Brief Title: Intracranial Genetically Modified Immune Cells (TGFβR2KO/IL13Rα2 CAR T-Cells) for the Treatment of Recurrent or Progressive Glioblastoma or Grade 3 or 4 IDH-Mutant Astrocytoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24717; NCI-2025-00342 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24717 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Astrocytoma, IDH-Mutant, Grade 3; Recurrent Astrocytoma, IDH-Mutant, Grade 4; Recurrent Glioblastoma
MeSH Terms: conditions — Astrocytoma; Lymphoma, Follicular; Glioblastoma | interventions — Specimen Handling; Immunotherapy, Adoptive; Fluorodeoxyglucose F18; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TGFβR2KO/IL13Rα2 CAR T-cells) (Experimental): Patients undergo leukapheresis and standard of care surgical resection with or without placement of Rickham catheter. Starting on day 0, patients receive autologous TGFβR2KO/IL13Rα2-CAR T cells intracranially over approximately 5 minutes QW. Cycles repeat weekly for up to 4 cycles (28 days) in the absence of disease progression or unacceptable toxicity. Patients may receive additional cycles if they continue to meet infusion criteria and have doses available for infusion. Patients also undergo CSF and blood sample collection and fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) and MRI throughout the study. Additionally, patients may undergo echocardiography at screening.
  Interventions: Procedure: Biospecimen Collection; Biological: Chimeric Antigen Receptor T-Cell Therapy; Procedure: Echocardiography; Other: Fludeoxyglucose F-18; Procedure: Intracranial Catheter Placement; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Resection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo CSF and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given autologous TGF-betaR2KO/IL13R-alpha2-CAR T cells intracranially
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Other: Fludeoxyglucose F-18 — Undergo FDG-PET
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Intracranial Catheter Placement — Undergo placement of Rickham catheter
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo FDG-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase I trial tests the safety, side effects and best dose of TGFβR2KO/IL13Rα2 chimeric antigen receptor (CAR) T-cells given within the skull (intracranial) in treating patients with glioblastoma or IDH-mutant grade 3 or 4 astrocytoma that has come back after a period of improvement (recurrent) or that is growing, spreading, or getting worse (progressive). CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack tumor cells. T cells are taken from a patient's blood. When the cells are taken from the patient's own blood, it is known as autologous. Then the gene for special receptors that bind to a certain proteins on the patient's tumor cells are added to the T cells in the laboratory. The special receptors are called CAR. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain tumors. Giving TGFβR2KO/IL13Rα2 CAR T cells may be safe, tolerable, and/or effective in treating patients with recurrent or progressive glioblastoma or grade 3 or 4 IDH-mutant astrocytoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety and determine the maximum tolerated dose (MTD) of intracranial (IC) administration of TGFβR2KO/IL13Rα2-CAR T cell therapy.

SECONDARY OBJECTIVES:

I. In participants who receive at least 50% of the assigned cell dose for each of the four cycles and at least 70% of the total cumulative dose for all cycles (1-4):

Ia. Estimate overall response rates (ORR) and complete response (CR) rate at 3, 6, 9-months; and Ib. Estimate overall survival (OS) at 9-months. II. Determine feasibility of IC administered TGFβR2KO/IL13Rα2-CAR T cell therapy as assessed by leukapheresis and manufacturing processes, including ability to meet the TGFβR2KO/IL13Rα2-CAR T cell dose and product release requirements; III. Determine the maximum feasible dose (MFD), as assessed by leukapheresis, manufacturing, toxicity, and response data.

EXPLORATORY OBJECTIVES:

I. Descriptively compare CAR T persistence in the cerebrospinal fluid (CSF) and the blood, cytokine dynamics, and response among patients treated on institutional review boards (IRBs) 24717 and 13384.

II. Profile cytokine levels and graphically evaluate cytokine levels over time and changes in the presence of cytokine release syndrome (CRS) toxicity (CSF, tumor cavity fluid [TCF], peripheral blood [PB]).

III. Describe CAR T cell and endogenous immune cell populations (CSF, TCF, PB). IV. Describe tumor and tumor micro-environment markers and their relationship to treatment outcomes.

V. For participants who undergo secondary resection(s) or autopsy on study:

Va. Evaluate CAR T cell persistence in the tumor micro-environment, location of the CAR T cells with respect to the injection site; and Vb. Evaluate changes in IL13Rα2 antigen expression levels pre and post CAR T cell therapy.

VI. Through the use of biomathematical modeling techniques, characterize tumor growth and its relationship to treatment outcomes.

OUTLINE: This is a dose-escalation study.

Patients undergo leukapheresis and standard of care surgical resection with or without placement of Rickham catheter. Starting on day 0, patients receive autologous TGFβR2KO/IL13Rα2-CAR T cells intracranially over approximately 5 minutes once weekly (QW). Cycles repeat weekly for up to 4 cycles (28 days) in the absence of disease progression or unacceptable toxicity. Patients may receive additional cycles if they continue to meet infusion criteria and have doses available for infusion. Patients also undergo CSF and blood sample collection and fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) and MRI throughout the study. Additionally, patients may undergo echocardiography at screening.

After completion of study treatment, patients are followed up on day 30, months 3, 6, 9 and 12, then yearly for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated main consent is processed. However, the research participant is allowed to proceed with surgery/Rickham placement and CAR T cell infusion only after the translated main consent form is signed
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies. If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Karnofsky performance status (KPS) ≥ 70%, Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy ≥ 4 weeks
* If the participant has a shunt, they must be informed of the following:

  * If the shunt is not programmable, the participant must be willing to have a programmable shunt placed prior to CAR T cell infusion, and
  * If the shunt is programmable, in order to proceed to the treatment portion of the study, the participant must be able to tolerate their shunt being functionally closed for at least 2 hours
* Participant has a prior histologically-confirmed diagnosis of a grade 3 or 4 IDH-mutant astrocytoma or glioblastoma, or has a prior histologically-confirmed diagnosis of a grade 2 or 3 astrocytoma and now has radiographic progression consistent with grade 3 or 4 IDH-mutant astrocytoma
* Relapsed disease: radiographic evidence of recurrence/progression of measurable disease after standard therapy, and ≥ 12 weeks after completion of front-line radiation therapy
* COH clinical pathology confirms IL13Rα2+ tumor expression by immunohistochemistry (H-score ≥ 80)
* No known contraindications to leukapheresis, steroids, or tocilizumab
* White blood cell (WBC) > 2000 /dl (or absolute neutrophil count [ANC] ≥ 1,000/mm^3) (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Platelets ≥ 75,000/mm^3 (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Hemoglobin ≥ 8g/dl (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Serum creatinine ≤ 1.6 mg/dL (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Oxygen (O2) saturation ≥ 95% on room air (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Seronegative for HIV antigen/antibody (Ag/Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative) (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test (to be performed within 14 days prior to leukapheresis unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Owing to higher frequency of wound-related complications, participants who require active bevacizumab therapy at the time of enrollment are excluded
* Participant has not yet recovered from toxicities of prior therapy
* Uncontrolled seizure activity and/or clinically evident progressive encephalopathy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Active autoimmune disease requiring systemic immunosuppressive therapy
* Active infection requiring intravenous (IV) antibiotics (e.g., minor scalp infection is not an exclusion)
* Known history of human immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Other active malignancy. Note: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2030-10-11 (Estimated); Study Completion 2030-10-11 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Up to 28 days
  Will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Rate and associated 90% Clopper and Pearson binomial confidence limits (90% CI) will be estimated for participants experiencing DLTs at the maximum tolerated dose schedule
Incidence of grade 3+ adverse events (AEs) | Up to 30 days after last dose of study drug
  Will be assessed using the CTCAE v 5.0. Tables will be created to summarize all toxicities and side effects by dose, time post treatment, organ, severity, attributions, and arm. In study participants who received the full schedule of 4 cycles.
Incidence of cytokine release syndrome | Up to 30 days after last dose of study drug
  Will be graded using American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Criteria. Tables will be created to summarize all toxicities and side effects by dose, time post treatment, organ, severity, attributions, and arm. In study participants who received the full schedule of 4 cycles.
Incidence of all other AEs | Up to 30 days after last dose of study drug
  Will be assessed using the CTCAE v 5.0. Neurotoxicity will be graded using ASTCT Consensus Criteria, Immune Effector Cell-Associated Hemophagocytic Lymphohistiocytosis-Like Syndrome grading system, and tumor inflammation-associated neurotoxicity grading system. Tables will be created to summarize all toxicities and side effects by dose, time post treatment, organ, severity, attributions, and arm.

SECONDARY OUTCOMES:
Overall response rate | At 3, 6, and 9 months
  Evaluated using Response Assessment in Neuro-Oncology (RANO) criteria. Will estimate the rates (90% CI) of disease response.
Complete response rate | At 3, 6, and 9 months
  Evaluated using RANO criteria. Will estimate the rates (90% CI) of disease response.
Overall survival (OS) | From cycle 1 to last contact or death from any cause, assessed at 9 months
  Will estimate the rates (90% CI) of OS. Kaplan Meier methods will be used to estimate median OS and graph the results.
Ability to meet the TGFβR2KO/IL13Rα2-CAR T cell dose requirements (product feasibility) | Up to 1 year
Ability to meet product release requirements (product feasibility) | Up to 1 year
Maximum feasible dose (MFD) | Up to 1 year
  The MFD will be determined based on observed toxicities/DLTs, including toxicities experienced in later cycles (5+), leukapheresis, manufacturing, and response data.

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Badie, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States